CLINICAL TRIAL: NCT05107297
Title: Comparison of National Early Warning Score (NEWS) & Sepsis Patient Evaluation in the Emergency Department (SPEED) for The Early Identification of Sepsis in the Emergency Department
Brief Title: Comparison to Early Detect of the Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Hassan Mostafa Abdellah, resident, Assiut University
Other Study IDs: sepsis identification
Record Dates: First submitted 2021-10-24; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Sepsis Scores

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to identify co-variates associated with 30-day mortality in septic patients admitted to the emergency department in order to improve morbidity & mortality as a sequence of sepsis in Assiut & Suez Canal Universities by comparing both scores by utilizing parameters that are readily available .

DETAILED DESCRIPTION:
There are a relatively large number of conditions where urgent intervention is required in order to secure the best outcome for the patient. Examples include sepsis, myocardial infarction (MI). Clinical diagnosis of some of these conditions is not always straightforward, but a common theme is that many present with deranged physiology and vital signs. Implementation of an early warning score on arrival at hospital has helped to identify seriously ill patients .

There is a high mortality rate associated with severe infection at all ages Sepsis occurs when life-threatening organ dysfunction is associated with infection.

What is a national early warning score (NEWS)? The following six simple physiological parameters are included in the scoring system: respiratory rate, oxygen saturation, temperature; the normal human body temperature range is typically stated as 36.5-37 °C( ), systolic blood pressure, pulse rate & level of consciousness.

What is a sepsis patient evaluation in the emergency department (SPEED)? The following simple clinical, physiological and laboratory parameters are included in the scoring system : hypotension (systolic pressure <90 mmHg) hypothermia (body temperature <36.0°C) , hypoxemia (pulse oximetry <90%), low hematocrit (hematocrit <0.38), Acidosis (blood PH < 7.35), elevated blood lactate >2.4 mmol/L & source of infection as pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 80 years.
* Patients of both genders.

Exclusion Criteria:

* Patient refusal .
* Accepts Healthy Volunteers .
* Aged below 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all gender entering the emergency deparment from 18 years to 80 years with no acceptance of healthy volunteers .
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Mortality . | 30 days
  Mortality during the 30 day follow-up.

SECONDARY OUTCOMES:
Hospital admission . | Day 0
  Admission to hospital from the Emergency Department.
ICU/HDU admission . | Day 0
  Admission to the Intensive Care Unit or High Dependency Unit from the Emergency Department .
Readmission in the ED . | Hour 72, Day 30
  Re-visits to the ED after the index-visit .

REFERENCES:
- [Background] Churpek MM, Snyder A, Han X, Sokol S, Pettit N, Howell MD, Edelson DP. Quick Sepsis-related Organ Failure Assessment, Systemic Inflammatory Response Syndrome, and Early Warning Scores for Detecting Clinical Deterioration in Infected Patients outside the Intensive Care Unit. Am J Respir Crit Care Med. 2017 Apr 1;195(7):906-911. doi: 10.1164/rccm.201604-0854OC. PMID 27649072
- [Background] Usman OA, Usman AA, Ward MA. Comparison of SIRS, qSOFA, and NEWS for the early identification of sepsis in the Emergency Department. Am J Emerg Med. 2019 Aug;37(8):1490-1497. doi: 10.1016/j.ajem.2018.10.058. Epub 2018 Nov 7. PMID 30470600
- [Background] Bewersdorf JP, Hautmann O, Kofink D, Abdul Khalil A, Zainal Abidin I, Loch A. The SPEED (sepsis patient evaluation in the emergency department) score: a risk stratification and outcome prediction tool. Eur J Emerg Med. 2017 Jun;24(3):170-175. doi: 10.1097/MEJ.0000000000000344. PMID 26524675